CLINICAL TRIAL: NCT06855849
Title: An Open-label, Single-arm, Multicenter Phase II Study to Evaluate the Efficacy of Amivantamab in Combination With FOLFIRI as a Second-line Treatment in Patients With RAS/BRAF Wild-type Advanced Colorectal Cancer Progressing on Prior Anti-EGFR Based Treatment.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-3346-002
Record Dates: First submitted 2025-02-24; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: RAS/BRAF Wild-type Advanced Colorectal Cancer Patients
MeSH Terms: interventions — amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amivantamab in combination with FOLFIRI (Experimental): Amivantamab will be administered as an IV infusion in 28-day cycles in combination with FOLFIRI IV infusion every 2 weeks.
  Interventions: Drug: Amivantamab + FOLFIRI

INTERVENTIONS:
Drug: Amivantamab + FOLFIRI — The dosage of amivantamab will be based on the participant's body weight during screening. Participants will receive 1,050 mg if BW is <80 kg or 1,400 mg if BW is ≥80 kg.
  * Cycle 1: once weekly (with the first dose split over Day -2 [350 mg, IVF for 4-6hrs] and Day -1 [remainder of the dose, IVF for 6-8hrs]; subsequent dose [planned dose IVF over 2 hrs]).
  * Cycles 2+: Days 1 and 15 of each cycle (planned dose IVF over 2 hrs) On days when both amivantamab and chemotherapy are administered, amivantamab should be administered before chemotherapy. In general, leucovorin 400 mg/m2 IV over 2 hours and irinotecan 180 mg/m2 IV over 90 min, then 5-FU 400 mg/m2 IV bolus followed by 5-FU continuous infusion 2,400 mg/m2 over approximately 46-48 hours or 1,200 mg/m2/day for two days. Irinotecan and leucovorin may be administered concurrently (via separate infusion lines) or sequentially according to the institutional standard.

SUMMARY:
This trial is a multicenter, single arm study of efficacy of amivantamab in combination with FOLFIRI in RAS/BRAF wild-type advanced colorectal cancer patients progressed prior treatment including oxaliplatin based chemotherapy. This trial will be conducted by Severance Hospital that is responsible for the project management of the trial. Patient recruitment will take at 3 institutions.

Participants will be treated for up to 24 cycles (approximately 2 years) after initiation of treatment with intravenous 1050mg(BW<80kg) or 1400mg(BW≥80kg) of amivantamab every 4 weeks in combination with FOLFIRI. FOLFIRI includes folic acid, 5-FU and irinotecan. FOLFIRI will be administered intravenously with folic acid 400 mg/m², 5-FU 2400 mg/m², and irinotecan 180 mg/m² every 2 weeks. This study will use ORR based on RECIST 1.1 criteria as the primary endpoint and the tumor assessment will be done every 8 weeks. Secondary endpoints are DCR, PFS, OS, and safeties. Exploratory biomarkers in tumor tissue and ctDNA in blood will be investigated in both pre-treatment and post-treatment periods.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥19 years of age.
2. The participant must have been previously diagnosed with histologically or cytologically confirmed unresectable or metastatic adenocarcinoma of the colon or rectum.
3. The participant must have a previously characterized tumor with wild-type KRAS, NRAS, and BRAF without evidence of ERBB2/HER2 amplification by immunohistochemistry (IHC) test. Local guidelines and SoC also require evaluation of dMMR/MSI-H status.
4. The participant must be diagnosed with CRC and should have received anti-EGFR and oxaliplatin-based systemic therapy in the metastatic setting (no more than one prior line of systemic therapy is allowed). According to local regulatory approvals and SoC guidelines, the participant must also be eligible for treatment with FOLFIRI.
5. Participants must have measurable disease according to RECIST v1.1. If only one measurable lesion exists, it may be used for the screening biopsy.
6. Participants must have ECOG PS 0 or 1.
7. Life expectancy ≥12 weeks as judged by the Investigator.
8. Participants must have adequate organ and bone marrow function as follows, without a history of red blood cell transfusion, platelet transfusion, or use of granulocyte colony-stimulating factor (G-CSF) within five days prior to the date of the laboratory test.

   A. Hemoglobin ≥ 8.0 g/dL B. Absolute neutrophil count ≥1.5ⅹ109/L C. Platelets ≥100ⅹ109/L D. ALT and aspartate aminotransferase (AST) ≤3ⅹupper limit of normal (ULN). If liver metastases are present, ≤ 5ⅹULN E. Total bilirubin ≤1.5ⅹULN (participants with Gilbert's syndrome can enroll if conjugated bilirubin is within normal limits) F. Serum creatinine ≤ 1.5ⅹULN, or calculated by Cockcroft-Gault formula (Refer to Appendix 9: Cockcroft-Graft Formula for Estimated Creatinine Clearance for formula) or directly measured creatinine clearance ≥ 50 mL/min
9. Negative serum pregnancy test within two weeks before the first study dose in all women of childbearing potential.
10. The subject and their partners must be willing to avoid pregnancy during the trial. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must be willing to use adequate contraception.
11. The participant must sign an ICF (or their legally acceptable representative must sign) indicating that he or she understands the purpose and procedures required for the study and is willing to participate.
12. Participants must be willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria:

1. Participants who have received prior irinotecan-based chemotherapy.
2. Participants with an identified mutation in KRAS, NRAS, BRAF, or ERBB2/HER2 amplification by immunohistochemistry (IHC) test.
3. Participant has an uncontrolled illness, including but not limited to the following:

   A. Active bleeding diathesis B. Impaired oxygenation requiring continuous oxygen supplementation C. Psychiatric illness/social situation that would limit compliance with study requirements.
4. Participants have known active CNS metastases or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least four weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable, and without requirement of steroid treatment for at least 14 days before the first dose of study treatment.
5. Participants with positive serology for HIV and HCV.

   A. Positive hepatitis C antibody (anti-HCV [hepatitis C virus]):

   Exception: Participants with a prior history of HCV who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
6. Anticancer treatment within 14 days before the start of trial treatment, e.g., cytoreductive therapy, radiotherapy (except for palliative bone-directed radiotherapy), immune therapy, or cytokine therapy.
7. Major surgery within 28 days before the start of trial treatment (excluding prior diagnostic biopsy).
8. Participants with a medical history of myocardial infarction within six months before treatment, symptomatic CHF (New York Heart Association Class II to IV), unstable angina pectoris, clinically significant cardiac arrhythmias, or a recent (< 6 months) cardiovascular event, including myocardial infarction, unstable angina pectoris, and stroke.
9. Gastrointestinal perforation, fistula, or any arterial thromboembolic event within six months, or any significant gastrointestinal bleeding or significant venous thromboembolism within three months prior to treatment (except for stable venous thromboembolism on ongoing appropriate anticoagulation treatment).
10. History of (non-infectious) ILD/pneumonitis, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within seven days before the first dose of the study drug.
12. Participants have a known previous or concurrent malignancy that has progressed or required active treatment within the past five years.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma or cervical cancer in situ) who have undergone potentially curative therapy are not excluded.
13. Toxicities from previous anticancer therapies should have resolved to baseline levels or Grade 1 or less prior to the first dose of study treatment (except for alopecia or post-radiation skin changes [any grade], and Grade ≤2 hypothyroidism stable on hormone replacement).
14. The participant has had prior chemotherapy or targeted cancer therapy with an investigational anticancer agent within two weeks or four half-lives, whichever is longer, before the first administration of the study drug.
15. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | every 8 weeks Up to 2 years 11 months
  Efficacy Analysis Set includes all patients who have received at least 1 dose of the study drug, had measurable disease at baseline according to RECIST 1.1, and had at least 1 post-baseline tumor response assessment. Patients with evidence of disease progression or death before the first scheduled assessment of tumor response will be included in this Analysis Set. It will be the primary analysis set for tumor response.
  Primary efficacy endpoints will be based upon investigators' tumor assessments per RECIST 1.1 and will be summarized as follows to evaluate the preliminary anticancer activities of amivantamab and FOLFIRI combination. Overall response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy by RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No